CLINICAL TRIAL: NCT00531921
Title: Correlation of Donor Proinflammatory mRNA Profiles With Early Outcomes of Thoracic and Abdominal Transplantation
Brief Title: Effects of Donor and Recipient Genetic Expression on Heart, Lung, Liver, or Kidney Transplant Survival
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-03
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Heart Transplantation; Kidney Transplantation; Liver Transplantation; Lung Transplantation
Keywords: Heart Diseases; Kidney Diseases; Liver Diseases; Liver Failure; Lung Diseases; Transplant; Transplantation, Homologous; Rejection; Kidney Failure
MeSH Terms: conditions — Heart Diseases; Kidney Diseases; Liver Diseases; Liver Failure; Lung Diseases; Rejection, Psychology; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples to evaluate the heart, kidney, liver, and lung
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Kidney transplants: patients from 5 specific sites
- Liver transplants: patients from 5 specific sites
- Heart transplants: patients from 5 specific sites
- Lung transplants: patients from 5 specific sites

SUMMARY:
Activity of genes in donor tissues that are involved in inflammation are thought to be involved with early organ dysfunction, increased immune responses in transplant recipients, and organ rejection. The purpose of this study is to determine the relationship between genetic expression in donor and recipient tissue with transplant survival. Participants in this study will have received heart, lung, liver, or kidney transplants.

DETAILED DESCRIPTION:
Inflammation and injuries to transplanted organs during the immediate post-operative period may be linked to early organ dysfunction and higher rates of transplant rejection in the recipient. Currently, mRNA expression of proinflammatory genes in donor tissues is thought to be a risk factor for early organ transplant dysfunction, increased expression of the recipients cell-mediated immunity genes, and organ rejection. The purpose of this study is to test the association between proinflammatory mRNA expression in donor samples and subsequent development of early organ dysfunction in kidney, lung, and liver transplant recipients. This study will also test the effects of proinflammatory mediators expressed in the transplanted organ pre- and post-reperfusion on organ rejection and genes expressed in cell mediated immune responses. This will be achieved by identifying the proinflammatory immune responses and their mechanisms.

This study will consist of up to 11 study visits over a period of 2 years. The baseline visit will occur 24 hours prior to organ transplantation. Follow-up visits will occur daily for Days 1 to 3 (for lung transplant recipients only) and on Day 7, Week 6, and Months 3, 6, 9, 12, 18, and 24 post-transplant. At the baseline visit, a physical exam, medical history, demographics, vital signs measurements, blood collection, and collection of donor tissue sample will occur. For most or all other study visits, medication and adverse events tracking and blood collection will occur. Depending on the transplant type, participants will undergo the following procedures:

* Heart: Participants will undergo a heart biopsy that is part of standard clinical care following a heart transplant. An echocardiogram and an electrocardiogram will occur at most visits.
* Kidney: Renal biopsies will be performed 1 hour after reperfusion at the time of surgery. Urine collection will occur at most visits.
* Liver: Liver biopsies will be performed at the time of procurement and within 1 hour of reperfusion.
* Lung: Participants will undergo bronchoalveolar lavage that is part of standard clinical care following a lung transplant. A chest x-ray, an arterial blood gas test, a pulmonary function test, and 6-minute walking test will occur at some visits.

ELIGIBILITY:
Inclusion Criteria for all participants:

* Received single lung, heart, kidney, or liver transplant
* Specimens of donor tissues have been collected
* Parent or guardian willing to provide informed consent, if applicable

Inclusion Criteria for Kidney or Liver Transplant Participants:

* 70 years old or younger

Inclusion Criteria for Heart or Lung Transplant Participants:

* Between 16 and 70 years old

Exclusion Criteria for All Participants:

* Previous solid organ transplant
* Need for combined organ transplant
* HIV or hepatitis C virus infection
* Recipient of an organ from a hepatitis C virus-infected donor
* Clinical evidence of systemic bacterial infection in the recipient at the time of transplantation
* Living donor transplant recipient of either a kidney, liver, or lung

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Transplant patients evaluated for the association between proinflammatory mRNA expression from donor samples and subsequent development of early organ dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Association between proinflammatory mRNA expression in donor samples and subsequent development of early organ dysfunction in the immediate period following transplantation | Within first 7 days after transplant
Association of mRNA expression of proinflammatory mediatros in the transplanted organ in the immediate pre and post-reperfusion period with subsequent incidence of acute rejection and expression of genes involved in cell mediated immunity | 12 months after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Shaked, MD, PhD, Principal Investigator — University of Pennsylvania Medical Center
Locations (5):
- United States (5):
  - Northwestern Memorial Hospital (kidney and liver), Chicago, Illinois
  - Cornell University Medical College (kidney), Ithaca, New York
  - Columbia University (lung and liver), New York, New York
  - University of Pennsylvania (heart, kidney, liver, lung), Philadelphia, Pennsylvania
  - University of Wisconsin (heart and lung), Madison, Wisconsin

REFERENCES:
- [Background] Fox-Marsh A, Harrison LC. Emerging evidence that molecules expressed by mammalian tissue grafts are recognized by the innate immune system. J Leukoc Biol. 2002 Mar;71(3):401-9. PMID 11867677
- [Background] Isobe M, Suzuki J. New approaches to the management of acute and chronic cardiac allograft rejection. Jpn Circ J. 1998 May;62(5):315-27. doi: 10.1253/jcj.62.315. PMID 9626898
- [Background] Jiang S, Lechler RI. CD4+CD25+ regulatory T-cell therapy for allergy, autoimmune disease and transplant rejection. Inflamm Allergy Drug Targets. 2006 Dec;5(4):239-42. doi: 10.2174/187152806779010981. PMID 17168794
- [Background] Kaplan B, Srinivas TR, Meier-Kriesche HU. Factors associated with long-term renal allograft survival. Ther Drug Monit. 2002 Feb;24(1):36-9. doi: 10.1097/00007691-200202000-00007. PMID 11805720
- [Background] Lande JD, Patil J, Li N, Berryman TR, King RA, Hertz MI. Novel insights into lung transplant rejection by microarray analysis. Proc Am Thorac Soc. 2007 Jan;4(1):44-51. doi: 10.1513/pats.200605-110JG. PMID 17202291
- [Background] Reding R, Gras J, Truong DQ, Wieers G, Latinne D. The immunological monitoring of alloreactive responses in liver transplant recipients: a review. Liver Transpl. 2006 Mar;12(3):373-83. doi: 10.1002/lt.20704. PMID 16498661
- [Background] Zheng XX, Sanchez-Fueyo A, Sho M, Domenig C, Sayegh MH, Strom TB. Favorably tipping the balance between cytopathic and regulatory T cells to create transplantation tolerance. Immunity. 2003 Oct;19(4):503-14. doi: 10.1016/s1074-7613(03)00259-0. PMID 14563315
- [Result] Cantu E, Lederer DJ, Meyer K, Milewski K, Suzuki Y, Shah RJ, Diamond JM, Meyer NJ, Tobias JW, Baldwin DA, Van Deerlin VM, Olthoff KM, Shaked A, Christie JD; CTOT Investigators. Gene set enrichment analysis identifies key innate immune pathways in primary graft dysfunction after lung transplantation. Am J Transplant. 2013 Jul;13(7):1898-904. doi: 10.1111/ajt.12283. Epub 2013 May 24. PMID 23710539
- [Derived] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- See also: Click here for the Clinical Trials in Organ Transplantation (CTOT) public Web site — http://www.ctotstudies.org